CLINICAL TRIAL: NCT06593873
Title: Effect of Preclinical Training in Periodontal Instrumentation on Undergraduate Students' Anxiety, Clinical Performance and Satisfaction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Okan University (Other)
Responsible Party: Principal Investigator, Sibel Kayaalti-Yuksek, Associate professor, Okan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2024/176
Record Dates: First submitted 2024-09-03; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Preclinical Education; Typodont-phantom Head; Anxiety
Keywords: Preclinical education; Typodont-phantom head; Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: This study included 60 fourth-year undergraduate students from Faculty of Dentistry, randomly divided into two groups. Both groups received one hour of theoretical periodontal training: the first, lasting 30 minutes, covered detailed instruction on comprehensive periodontal examination and supragingival instrumentation process through a multimedia presentation, and the second, also 30 minutes, demonstrated practical aspects (working area, support techniques, and positioning) on a patient. Group 1 received theoretical training, while Group 2 had the theoretical plus 60 minutes of preclinical practical training using a typodont-phantom head with artificial calculus. Immediately before performing supragingival instrumentation on their first patients, students completed a state anxiety test. After the procedures, participants completed VAS to rate training satisfaction. The student's clinical performance was evaluated using the scaling operation score sheet.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1: Theoretical training only (Control Group) (Other): Group 1 (control group) will receive only theoretical training.
  Interventions: Other: Theoretical periodontal education
- Group 2: Theoretical training+ Preclinical practical training with typodont-phantom head(Test group) (Other): Group 2 (test group) will receive training with typodont-fantom head in addition to theoretical training.
  Interventions: Other: Use of typodont head model in addition to theoretical periodontal education

INTERVENTIONS:
Other: Use of typodont head model in addition to theoretical periodontal education — Use of typodont phantom head model in addition to theoretical periodontal education
  Arms: Group 2: Theoretical training+ Preclinical practical training with typodont-phantom head(Test group)
Other: Theoretical periodontal education — Theoretical periodontal training only
  Arms: Group 1: Theoretical training only (Control Group)

SUMMARY:
The purpose of this study was to evaluate the effect of periodontal instrumentation preclinical training using a teaching typodont-phantom head model on undergraduate students; anxiety levels, clinical performance, and educational satisfaction.

DETAILED DESCRIPTION:
Sixty fourth-year undergraduate dental students will be randomly divided into two groups. Both groups will receive one hour of theoretical periodontal training.

Group 1 will receive only theoretical training, while Group 2 will complete this training as well as pre-clinical practical training with a typodont-phantom head with synthetic calculus. Before performing supragingival instrumentation on their first patient, students in both groups will be administered a state anxiety test. After the procedures, participants will complete a Visual Analog Scale (VAS) to assess training satisfaction. Students' clinical performance will be evaluated using the scaling procedure score sheet.

ELIGIBILITY:
Inclusion Criteria:

* To be a fourth year student of the Faculty of Dentistry
* To successfully complete pre-clinical theoretical and practical training
* To perform periodontal treatment for the first time in the undergraduate clinic

Exclusion Criteria:

* Not being a fourth year student of the Faculty of Dentistry
* Lack of attendance to pre-clinical theoretical training
* Failure to demonstrate competence in pre-clinical theoretical education
* Having previously performed periodontal treatment in undergraduate clinic

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Comparison of state anxiety scores of the participants | baseline
  After completing training, students in both groups took a state anxiety test using the State-Trait Anxiety Inventory (STAI) before performing supragingival instrumentation. The STAI, which assesses current anxiety levels with 20 items, provides a total score from 20 to 80 points.The STAI was completed using a 4-point Likert scale for each question. Items 3, 4, 6, 7, 9, 12, 13, 14, 17, and 18 contribute positive scores, which increased the total anxiety score. Conversely, items 1, 2, 5, 8, 10, 11, 15, 16, 19, and 20 contributed negative scores, which decreased the total anxiety score. Each item was scored between 1 (or -1) and 4 (or -4) based on its positive or negative nature, and a constant of 50 is added to the total score. Higher scores indicated higher levels of state anxiety.
Comparison of scaling operation scores among study groups | baseline
  The clinical performance of the participants was evaluated by a blind periodontologist using a scaling operation score sheet.The scale assessed clinical performance across four categories: preoperative preparation, intraoperative operation, periodontal probing, and supragingival instrumentation. Each category included specific criteria with assigned points, resulting in a maximum score of 100. The evaluation focused on fundamental aspects including equipment preparation, positioning, probing techniques, and supragingival scaling.

SECONDARY OUTCOMES:
Evaluating participants' satisfaction levels | baseline
  The evaluation of students' satisfaction with their training following the intervention was conducted using a Visual Analog Scale (VAS). The VAS was presented as a horizontal line, 10 centimeters in length, with endpoints labeled to represent the extremes of satisfaction. One end of the line was labeled 0 to represent very low satisfaction, and the other end was labeled 10 to represent very high satisfaction. Participants marked a point on the line that best reflected their level of satisfaction. The distance from the 0 end to the participant's mark was measured in millimeters, providing a quantitative score of their satisfaction level.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Istanbul Okan Universitiy, Istanbul
  - Sibel Kayaaltı Yüksek, Istanbul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kayaalti-Yuksek S, Besiroglu-Turgut E, Agirman M, Keles GC. Effect of preclinical training in periodontal instrumentation on undergraduate students' anxiety, clinical performance, satisfaction. BMC Oral Health. 2025 Jul 15;25(1):1167. doi: 10.1186/s12903-025-06041-y. PMID 40665307